CLINICAL TRIAL: NCT04347720
Title: Relative Effectiveness and Safety of Pharmacotherapeutic Agents for Patent Ductus Arteriosus (PDA) in Preterm Infants: A National Comparative Effectiveness Research (CER) Project
Brief Title: Canadian National PDA Treatment Study
Acronym: CANRxPDA
Status: Completed | Type: Observational
Sponsor: IWK Health Centre (Other)
Collaborators: Provincial Health Services Authority British Columbia (Other); Children's Hospital of Eastern Ontario (Other); CHU de Quebec-Universite Laval (Other); Foothills Medical Centre (Other); Victoria General Hospital (Unknown); The Hospital for Sick Children (Other); Health Sciences Centre, Winnipeg, Manitoba (Other); St. Justine's Hospital (Other); Queen's University (Other); MOUNT SINAI HOSPITAL (Other); Royal Alexandra Hospital (Other); Regina General Hospital (Other); Royal University Hospital Foundation (Other); St. Boniface Hospital (Other); The Moncton Hospital (Unknown); Horizon Health Network (Other); Sunnybrook Health Sciences Centre (Other); Windsor Regional Hospital (Other); Royal Columbian Hospital Foundation (Other); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other); London Health Sciences Centre (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Souvik Mitra, MD MSc FRCPC, Assistant Professor, IWK Health Centre
Other Study IDs: 1025627
Record Dates: First submitted 2020-04-12; First posted 2020-04-15 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Patent Ductus Arteriosus; Extreme Prematurity
Keywords: indomethacin; ibuprofen; acetaminophen
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Indomethacin; Ibuprofen; Acetaminophen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Indomethacin Arm: Intravenous indomethacin at 0.1-0.3 mg/kg IV every 12-24h for a total of 3 doses as choice of initial pharmacotherapy.
  Interventions: Drug: Indomethacin
- Standard dose ibuprofen Arm: Standard dose ibuprofen [Oral/intravenous] at 10 mg/kg followed by 2 doses of 5mg/kg at 24 h intervals irrespective of postnatal age as choice of initial pharmacotherapy.
  Interventions: Drug: Ibuprofen
- Adjustable dose ibuprofen Arm: Adjustable dose ibuprofen [Oral/intravenous] as choice of initial pharmacotherapy. The dose of ibuprofen will be 10 mg/kg followed by 2 doses of 5 mg/kg at 24 h intervals if treated within the first 7 days after birth. Higher doses of ibuprofen up to 20 mg/kg followed by 2 doses of 10 mg/kg at 24 h intervals if treated after the postnatal age cut-off for lower dose as per the local center policy
  Interventions: Drug: Ibuprofen
- Acetaminophen Arm: Acetaminophen [Oral/intravenous] at 15mg/kg every 6h for 3-7 days as choice of initial pharmacotherapy.
  Interventions: Drug: Acetaminophen
- Control group: Infants <29 weeks GA with echocardiography-confirmed PDA but never received any pharmacotherapy
- Reference group: Infants <29 weeks GA who were never diagnosed with PDA

INTERVENTIONS:
Drug: Indomethacin — Intravenous formulation
  Other Names: indocid
  Groups: Indomethacin Arm
Drug: Ibuprofen — Intravenous and oral formulations
  Other Names: Advil; NeoProfen
  Groups: Adjustable dose ibuprofen Arm; Standard dose ibuprofen Arm
Drug: Acetaminophen — Intravenous and oral formulations
  Other Names: paracetamol
  Groups: Acetaminophen Arm

SUMMARY:
Patent ductus arteriosus (PDA) is the most common cardiovascular problem that develops in preterm infants. Persistent PDA may result in higher rates of death, chronic lung disease (CLD), pulmonary hemorrhage, necrotizing enterocolitis (NEC), acute kidney injury (AKI), intraventricular hemorrhage (IVH) and cerebral palsy. Currently available options to treat a PDA include indomethacin, ibuprofen or acetaminophen followed by surgical or interventional closure of the PDA if medical therapy fails.

Wide variation exists in PDA treatment practices across Canada. A survey conducted through the Canadian Neonatal Network (CNN) in 2019 showed that the most common choice of initial pharmacotherapy is standard dose ibuprofen. In view of the high pharmacotherapy failure rate with standard dose ibuprofen, there is a growing use of higher doses of ibuprofen with increasing postnatal age (with 32% of respondents currently adopting this practice) in spite of the fact that effectiveness and safety of higher ibuprofen doses have not been established in extremely preterm infants [<29 weeks gestational age (GA)]. In view of this large practice variation across Canadian neonatal intensive care units (NICUs), we are planning a comparative effectiveness study of the different primary pharmacotherapeutic agents used to treat the PDA in preterm infants.

Aims Primary: To compare the primary pharmacotherapeutic practices for PDA closure and evaluate their impact on clinical outcomes in extremely preterm infants (<29 weeks GA) Secondary: To understand the relevance of pharmacotherapeutic PDA treatment with respect to clinical outcomes in the real world.

Methods:

Participants: Extremely preterm infants (<29 weeks gestational age) with an echocardiography confirmed PDA who will be treated according to attending team

Interventions:

1. Standard dose ibuprofen [10-5-5 regimen, i.e., 10mg/kg followed by 2 doses of 5mg/kg at 24h intervals]
2. Adjustable dose ibuprofen [10-5-5 regimen if treated within the first week. Higher doses of ibuprofen up to a 20-10-10 regimen if treated after the postnatal age cut-off for lower dose as per the local center policy]
3. Intravenous indomethacin [0.1-0.3mg/kg every 12-24h for a total of 3 doses].
4. Acetaminophen [Oral/intravenous] (15mg/kg every 6h) for 3-7 days

Outcomes:

Primary: Failure of primary pharmacotherapy (Need for further medical and/or surgical/interventional treatment following an initial course of pharmacotherapy).

Secondary: (a) Receipt of 2nd course of pharmacotherapy; (b) Surgical/interventional PDA closure; (c) CLD (d) NEC (stage 2 or greater) (e) Severe IVH (Grade III-IV) (f) Definite sepsis (g) Stage 1 or greater AKI; (h) Post-treatment serum bilirubin; (i) Phototherapy duration; (j) All-cause mortality during hospital stay.

DETAILED DESCRIPTION:
In this study, we intend to generate real-world evidence (RWE) by analyzing real-world data (RWD) (defined as data generated during routine clinical practice) from a registry-based Comparative Effectiveness Research study.

The Canadian Neonatal Network (CNN) is a well-established patient registry that includes members from 31 hospitals and 17 universities across Canada. The Network maintains a standardized NICU database and provides a unique opportunity for researchers to participate in collaborative projects. We will use the principles of Hypotheses Evaluating Treatment Effectiveness (HETE) research, which are designed to evaluate the presence or absence of a pre-specified effect and/or its magnitude. The network has recent experience in conducting such a study where one CIHR-funded study to evaluate effectiveness of two modes of non-invasive ventilation in preterm infants is already underway in 20 NICUs across Canada.

The CNN's coordinating facility is located within the Maternal-Infant Care (MiCare) Research Center, Lunenfeld-Tanenbaum Research Institute (LTRI) at Mount Sinai Hospital (Toronto). Each participating site has highly trained abstractors who enter data from patient charts into the CNN database. The abstractors will also enter data specific to our project, which will allow us to obtain real-world data at a minimal cost with easy access to investigators for troubleshooting.

Statistical Analysis overview: Since the proposed study is a CER using RWD, we will examine and account for potential confounders at the analyses stage. As recommended for HETE studies using RWD, accuracy of results will be checked by performing complementary sensitivity analyses. The analyses will be conducted in 2 stages: unit-level protocol effectiveness analysis and a secondary drug-dosage effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* Extremely preterm infants (<29 weeks gestational age) with an echocardiography confirmed PDA who will be treated according to attending team

Exclusion Criteria:

* Any infant who received pharmacotherapy for a clinically symptomatic PDA without prior echocardiographic confirmation of the presence of PDA will be excluded from all analyses.

Max Age: 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants born less than 29 weeks of gestation admitted to the participating sites will be included in the study. The population of interest will be those preterm infants <29 weeks gestational age (including outborns) with echocardiography confirmed PDA who will be treated according to attending team. Infants <29 weeks GA with echocardiography-confirmed PDA but never received treatment will be included as the control population. Infants <29 weeks GA who were never diagnosed with PDA will be included as the reference population
Sampling Method: Probability Sample
Enrollment: 1663 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Failure of primary pharmacotherapy | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  Receipt of further medical and/or surgical/interventional treatment following an initial course of pharmacotherapy

SECONDARY OUTCOMES:
Receipt of 2nd course of pharmacotherapy | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
Surgical/interventional PDA closure | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
Chronic lung disease | birth through 36 weeks post menstrual age
  Oxygen or respiratory support requirement at 36 weeks' postmenstrual age or at discharge
Necrotizing enterocolitis | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  Stage 2 or greater as per Bell's criteria
Severe intraventricular hemorrhage | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  Grade III-IV according to Papile Criteria
Definite sepsis | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  Clinical symptoms and signs of sepsis and a positive bacterial culture in a specimen obtained from normally sterile fluids or tissue obtained at postmortem
Acute Kidney Injury | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)
  Stage 1 or greater according to the Neonatal AKI KDIGO classification
Post-treatment serum bilirubin | within 7 days of initiation of pharmacotherapy
Maximum serum AST and ALT (u/L) during treatment or within 1 week of treatment completion | within 7 days of completion of pharmacotherapy
All-cause mortality during hospital stay | through hospital discharge (approximately 20 weeks postnatal age unless death occurs first)

CONTACTS AND LOCATIONS:
Overall Officials: Souvik Mitra, MD, MSc, Principal Investigator — IWK Health Center, Halifax, Canada; Amish Jain, MBBS, PhD, Principal Investigator — Mount Sinai Hospital, Canada; Prakeshkumar Shah, MD, FRCPC, Principal Investigator — Mount Sinai Hospital, Canada
Locations (22):
- Canada (22):
  - Foothills Medical Centre, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - British Columbia Women's Hospital, Vancouver, British Columbia
  - Victoria General Hospital, Victoria, British Columbia
  - Health Sciences Centre, Winnipeg, Manitoba
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - IWK Health Center, Halifax, Nova Scotia
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Windsor Regional Hospital, Windsor, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Regina General Hospital, Regina, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Mitra S, Jain A, Ting JY, Ben Fadel N, Drolet C, Abou Mehrem A, Soraisham A, Jasani B, Louis D, Lapointe A, Dorling J, Khurshid F, Hyderi A, Kumaran K, Bodani J, Weisz D, Alvaro R, Adie M, Stavel M, Morin A, Bhattacharya S, Kanungo J, Canning R, Ye XY, Hatfield T, Gardner CE, Shah P. Relative effectiveness and safety of pharmacotherapeutic agents for patent ductus arteriosus (PDA) in preterm infants: a protocol for a multicentre comparative effectiveness study (CANRxPDA). BMJ Open. 2021 May 5;11(5):e050682. doi: 10.1136/bmjopen-2021-050682. PMID 33952559
- See also: Project funding information on the Canadian Institutes of Health Research (CIHR) Funding Decision Database — http://webapps.cihr-irsc.gc.ca/decisions/p/project_details.html?applId=410247&lang=en